CLINICAL TRIAL: NCT02671513
Title: A Tolerability and Pharmacokinetics Phase 1 Study of SHR6390 in Advanced Melanoma Patients
Brief Title: A Tolerability and Pharmacokinetics Study of SHR6390 in Advanced Melanoma Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR6390-I-102
Record Dates: First submitted 2016-01-24; First posted 2016-02-02 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-01

CONDITIONS: Melanoma
Keywords: Melanoma; Cycline-Dependent Kinase
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SHR6390 (Experimental): Each subject will receive a single dose of SHR6390 and then repeat doses following a 3 week/1 week off regimen.
  Interventions: Drug: SHR6390

INTERVENTIONS:
Drug: SHR6390 — SHR6390 either 50mg,75mg,100mg,125mg,150mg,175mg given orally, QD

SUMMARY:
SHR6390 is a small molecular,oral potent, selective CDK4/6 inhibitor. The purpose of this study is to investigate the safety/tolerability and the pharmacokinetic profile of SHR6390 in Chinese advanced melanoma patients by using a "3+3" dose escalation.Preliminary efficacy will be also investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed melanoma
* Unresectable stage III or IV melanoma patient
* companion with cell cycle pathway abnormal (e.g CDK4 amplify and/or CCND1 amplify and/or CDKN2A loss)
* Eastern Cooperative Oncology Group (ECOG) performance status:0-1
* Life expectancy ≥ 3 months
* Adequate function of major organs, meaning the following criteria should be met within 14 days before randomization:

Hemoglobin > 100g/L Neutrophils > 2.0×10^9/L Platelets > 100×10^9/L Total bilirubin < 1.5×the upper limit of normal (ULN) ALT and AST ≤ 1.5×ULN (≤ 5×ULN, if existing liver metastases) Creatinine ≤ 1 ULN Left ventricular ejection fraction (LVEF) ≥ 50% QTcF(Fridericia correction) male≤450 ms, female≤470 ms

* Good compliance of patient by physician's judgement
* Signed and dated informed consent

Exclusion Criteria:

* Previously received therapy of anti-tumor agent targeting at CDK4/6
* Less than 3 weeks from the last cell-toxicity chemotherapy, less than 6 weeks from last mitomycin or nitrosamine therapy
* Less than 3 weeks from any other anti-tumor therapy (including targets therapy, immunotherapy or other approved therapy)
* Having joined in other clinical trials within 4 weeks
* Uncontrolled/untreated brain metastasis (well-controlled/well-treated brain metastasis by physician's judgement is allowed)
* existing abnormal CTCAE≥grade 2 resulted from previous treatment
* uncontrollable symptomatic pleural effusion or ascites or require clinical intervention
* require continous treatment by steroids
* Factors influencing the usage of oral administration (e.g. unable to swallow, chronic diarrhea and intestinal obstruction, etc.)
* existing uncontrollable hypokalemia or hypomagnesemia
* history of serious allergy events or known being allergy constitution
* active HBV or HCV infection (HBV virus≥10e4 copies/ml, HCV virus≥10e3 copies/ml)
* History of immunodeficiency, acquired or congenital immunodeficiency, history of organ transplantation
* history of cardiac dysfunction, include(1)angina (2)clinical significant arrythmia or require drug intervention (3)myocardial infarction (4)heart failure (5) other cardiac dysfunction (judged by the physician); any cardiac or nephric abnormal ≥grade 2 found in screening
* Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test
* childbearing female who refuse to accept any contraception practice
* determined by the physician, any coexisting disease might lead to life threatening complications or avoid the patients from accomplishing the treatment(e.g serious hypertension, diabetes, thyroid dysfunction,etc.)
* history of neuropathy or dysphrenia, including epilepsy and dementia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-11 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 3 weeks
  The maximum-tolerated dose (MTD) will be defined as the maximum dose level at which no more than one out of three subjects experience a dose-limiting toxicity (DLT) within the first 3 week of the first cycle of multiple dosing.

SECONDARY OUTCOMES:
Evaluation of pharmacokinetic parameter of SHR6390: Cmax | 6 weeks
Evaluation of pharmacokinetic parameter of SHR6390: Tmax | 6 weeks
Evaluation of pharmacokinetic parameter of SHR6390: t1/2 | 6 weeks
Evaluation of pharmacokinetic parameter of SHR6390: AUC | 6 weeks
Number of patients experience adverse events | 6 months
objective response rate | every 8 weeks, up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, M.D, Principal Investigator — Beijing Cancer hospital,Peking University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No